CLINICAL TRIAL: NCT06556498
Title: Progrip Versus ProFlor: Two Fixation Free Devices for Laparoscopic Inguinal Hernia Repair: A Randomized Clinical Trial: The ProPro Study
Brief Title: Progrip Versus ProFlor: Two Fixation Free Devices for Laparoscopic Inguinal Hernia Repair
Acronym: ProPro
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, Full Professor of Surgery, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProPro study
Record Dates: First submitted 2024-06-29; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Hernia, Inguinal; Laparoscopic Surgery
Keywords: hernia surgery; inguinal hernia; fixation free repair; TAPP; laparoscopic surgery
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: we use progrip mesh and proflor mesh in different arms of patients
Masking Description: Compared progrip mesh with proflor mesh
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ProFlor group (Active Comparator): patients underwent to laparoscopic hernia repair with the use of ProFlor mesh
  Interventions: Procedure: Proflor group
- Progrip group (Active Comparator): patients underwent to laparoscopic hernia repair with the use of Progrip mesh
  Interventions: Procedure: Progrip group

INTERVENTIONS:
Procedure: Proflor group — evaluate the surgical outcomes of patients underwent to laparoscopic inguinal hernia repair with Proflor mesh.
  Arms: ProFlor group
Procedure: Progrip group — evaluate the surgical outcomes of patients underwent to laparoscopic inguinal hernia repair with Progrip mesh.
  Arms: Progrip group

SUMMARY:
there are currently two methods for fixation free laparoscopic inguinal hernia repair specifically based on the intrinsic properties of the device used. The Progrip mesh technique leaves the hernia orifice patent and relies on the established principle of strengthening the groin through scar tissue incorporation induced by foreign body reaction. In contrast, the ProFlor concept introduces a 3D dynamic regenerative scaffold that permanently obliterates the defect and regenerates the herniated inguinal barrier. This report presents the outcomes of laparoscopic techniques employing Progrip and ProFlor in randomized clinical trial. The results of this clinical study may have the potential to pave the way for innovative advancements in hernia repair techniques.

ELIGIBILITY:
Inclusion Criteria:

* bilateral inguinal hernia

Exclusion Criteria:

* Recurrent inguinal hernia
* Incarcerated inguinal hernia
* Hernia not in the inguinal area
* Signs of obvious local or systemic infection
* ASA score > 4
* Presenting with unstable angina or NYHA class of IV
* Pregnant
* Active drug user
* Immunosuppression, chemotherapy
* Chronic renal insufficiency
* Abdominal ascites
* Infection in area of the surgical field
* BMI >34

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative adverse events | 30-postoperative days
  postoperative adverse events. The primary objective of these evaluations was to detect any possible complications that may have arisen, including but not limited to recurrence, hematoma, seroma, testicular swelling, wound infection/abscesses, prosthesis displacement, or any other complication. We used clinical observation and radiological findings to detect these complications.

SECONDARY OUTCOMES:
Visual analogue score (VAS) | 1 - 6- 12 and 24 months
  The secondary endpoints included evaluations of postoperative pain. During follow-up control, patients were tasked with completing questionnaires aimed at evaluating their clinical conditions. To assess pain levels during the early stage (until four weeks postop.), the Visual Analogue Score (VAS) was employed. The VAS score is a widely recognized tool that enables patients to rate their pain on a scale from 0 to 10, where 0 signifies no pain and 10 indicates the most severe pain imaginable.
Carolinas Comfort Scale (CCS) | 1 - 6- 12 and 24 months
  The secondary endpoints included evaluations of discomfort and quality of life. During follow-up control, patients were tasked with completing questionnaires aimed at evaluating their clinical conditions. For long-term clinical evaluation starting from four weeks postop, patients were instructed to fill out the Carolinas Comfort Scale questionnaire (CCS), regarded as the optimal scoring system for discomfort, and other postoperative symptoms. The CCS questionnaire offered a more thorough insight into the patient's experience and facilitated the evaluation of their long-term outcomes.
  The CCS is a 23-itemquestionnaire that quantifies the severity of pain, mesh sensation, and movement limitation from the hernia or surgical site during the following 8 activities: lying down, bending over, sitting up, activities of daily living, coughing or deep breathing (Min. 0 with no discomfort in all activity; Max. 115 with maximum discomfort in all activity)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Di Buono, Principal Investigator — University of Palermo; Antoninoq Agrusa, Study Director — University of Palermo
Locations (1):
- Italy, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Buono G, Romano G, Rodolico V, Amato G, Zanghi G, Romano G, Calo PG, Agrusa A. Progrip versus ProFlor: two fixation-free devices for laparoscopic inguinal hernia repair-the Pro/Pro study, a randomized clinical trial. Surg Endosc. 2025 May;39(5):3113-3126. doi: 10.1007/s00464-025-11680-x. Epub 2025 Apr 1. PMID 40167608